CLINICAL TRIAL: NCT04722094
Title: Prevalence of Periodontitis in Patients With Plaque Psoriasis. A Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Researcher, University of Siena
Other Study IDs: PSO001
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis; Plaque Psoriasis; Periodontal Diseases; Periodontitis
MeSH Terms: conditions — Psoriasis; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva sample for miRNAs extraction (miRNAs 146a, 155, 223, 21)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Psoriasis: All patients pertaining to the Unit of Dermatology and affected by psoriasis will be screened for the inclusion in the study
  Interventions: Diagnostic Test: Full periodontal chart; Other: Saliva sampling

INTERVENTIONS:
Diagnostic Test: Full periodontal chart — A full periodontal chart will be carried out including all biometric periodontal variables: Probing Pocket Depth (PPD), Bleeding on Probing (BoP), presence of Plaque, recession (REC), Full Mouth Plaque Score (FMPS), Full Mouth Bleeding Score (FMBS), presence of furcation and mobility. Periodontal status, as assessed by the periodontal chart, will be evaluated following the New Classification of Periodontal and Peri implant diseases.
Other: Saliva sampling — Saliva samples for miRNAs detection will be taken before starting the visit.

SUMMARY:
Psoriasis is a chronic inflammatory disease with a multi-factorial etiology which affects the epidermis and dermis. It affects around 1-3% of the general population and its most frequent form is plaque psoriasis (around 80-90% of the overall psoriasis cases). Psoriasis severity and extension are usually measured through 2 scores: Psoriasis Area Severity Index (PASI) and Body Surface Area (BSA). Periodontitis is a chronic inflammatory disease mediated by the biofilm and with a multi-factorial etiology. Its manifestation entails the destruction of the periodontal tissues surrounding the teeth; the final stage of disease is characterised by tooth loss. Periodontitis severity and extension are usually evaluated through surrogate variables such as: BoP (Bleeding on Probing), PPD (Probing Pocket Depth) e REC (Recession). Both diseases present overlapping genetic and pathophysiologic features, as well as common risk factors (e.g. genetic polymorphisms, smoking habit, obesity, diabetes etc.).

miRNAs are small non-coding molecules involved in the regulation of various biologic processes thanks to their interaction with mRNAs. Active inflammatory processes either in the oral cavity or at a systemic level tend to alter the concentration of salivary miRNAs. No study so far has ever profiled the levels of specific salivary miRNAs in patients with psoriasis and periodontitis.

Some case-control studies highlighted a higher prevalence of periodontitis in patients with psoriasis when compared to healthy controls. Nonetheless, epidemiological data regarding periodontitis prevalence in patients with psoriasis are lacking; moreover, few data are available regarding the relationship between the severity of psoriasis and the severity of periodontitis, together with the effect of common risk factors (e.g. diet, obesity, physical activity, sleep quality etc.).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Diagnosis of plaque psoriasis
* Ability and willingness to give informed consent

Exclusion Criteria:

* Inability of unwillingness to give informed consent
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by Plaque Psoriasis and meeting the inclusion criteria will be screened for the inclusion in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-06-25 (Estimated); Study Completion 2021-08-25 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Periodontitis in patients with Plaque psoriasis | Baseline
  The prevalence of patients with a diagnosis of periodontitis among the included cohort will be measured.

SECONDARY OUTCOMES:
relationship between salivary miRNAs concentration and the severity of psoriasis and periodontitis | Baseline
  salivary levels of miRNAs will be related to the severity of psoriasis and periodontitis

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Discepoli, DDS, MsC, PhD, Principal Investigator — University of Siena
Locations (1):
- AOUS, Siena, Italy

IPD SHARING:
Plan to Share IPD: No